CLINICAL TRIAL: NCT07152197
Title: Effects of a Resistance Exercise Training Program on Skeletal Muscle Quality, Functional Capacity, and Quality of Life in Young Individuals With and Without Hereditary Sensorimotor Polyneuropathy
Brief Title: Effects of Resistance Exercises in Hereditary Sensory-Motor Neuropathy (Charcot-Marie-Tooth Disease)
Acronym: PNP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de La Frontera (Other)
Responsible Party: Principal Investigator, Fernando Javier Valenzuela Aedo, Clinical Professor, Universidad de La Frontera
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 054/25
Record Dates: First submitted 2025-08-18; First posted 2025-09-03 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Polyneuropathy; Charcot Marie Tooth Disease (CMT)
Keywords: Charcot Marie Tooth Disease (CMT); Resistance Training; Muscle Quality; Quality of Life
MeSH Terms: conditions — Polyneuropathies; Charcot-Marie-Tooth Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The expert evaluators of the pre- and post-intervention variables will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Charcot Marie Tooth (CMT Group) (Experimental): Participants with Charcot-Marie-Tooth (CMT) will perform an 8-week supervised lower limb Progressive Resistance Exercise Training (RET) program, 3 times per week. Assessments will be conducted pre- and post-intervention to evaluate muscle quality, functional capacity, and quality of life.
  Interventions: Other: Progressive Resistance Exercise Training
- CONTROL Group (Active Comparator): Healthy participants (without Charcot Marie Tooth) will perform an 8-week supervised lower limb Progressive Resistance Exercise Training (RET) program, 3 times per week. Assessments will be conducted pre- and post-intervention to evaluate muscle quality, functional capacity, and quality of life.
  Interventions: Other: Progressive Resistance Exercise Training

INTERVENTIONS:
Other: Progressive Resistance Exercise Training — Progressive Resistance Exercise Training Supervised (RET) focusing on lower limbs. Warm-up (5 min cycling), followed by 5 sets of leg press, leg extension, leg curl, and weighted dorsiflexion. Cool-down with flexibility exercises. Load progression from 60% to 80% of 1Repetition Maximum across 8 weeks. Participants must complete ≥80% of sessions. Evaluators of pre- and post-intervention outcomes will be blinded.

SUMMARY:
The goal of this clinical trial is to compare the effects of an 8-week resistance exercise training program on skeletal muscle quality, functional capacity, and quality of life in young individuals aged 15 to 29 years, with and without Hereditary Sensorimotor Polyneuropathy (HSPN).

The main questions to answer are:

What is the effect of an 8-week resistance exercise training program on skeletal muscle quality, functional capacity, and quality of life in young individuals with and without HSPN?

Will the percentage of improvement after the program be greater in participants with HSPN compared to those without, due to greater baseline alterations?

Researchers will compare the resistance exercise training program with baseline conditions to determine its effectiveness in improving skeletal muscle quality, functional capacity, and quality of life.

Participants will undergo a supervised lower-limb resistance exercise program (3x/week) for 8 weeks. The intervention will include progressive loads from 60% to 80% of 1-Repetition Maximum (1RM), with exercises targeting the major lower limb muscle groups. All participants will complete pre- and post-intervention evaluations, including ultrasound assessment of muscle architecture, functional capacity tests, strength measurements, body composition analysis, and quality of life questionnaires.

DETAILED DESCRIPTION:
Introduction: Hereditary sensorimotor polyneuropathy (HSPN), also known as Charcot-Marie-Tooth disease (CMT), is the most prevalent group of hereditary neuromuscular disorders. It is characterized by muscle distal weakness, muscle atrophy, sensory loss, balance impairments, skeletal deformities and, in some cases, respiratory dysfunction. These impairments lead to reduced muscle quality, functional capacity, and quality of life. Muscle quality encompasses both morphological and functional aspects of skeletal muscle, including muscle architecture, composition, and strength.

Resistance exercise training (RET) has been shown to improve strength, muscle morphology, and functional performance in various populations. However, there is limited evidence on its effectiveness in individuals with HSPN, particularly in young adults. No studies to date have compared the effects of lower-limb-focused RET on muscle quality, functional capacity, and quality of life in young adults with and without HSPN.

Objectives:

The primary objetive of this study will be to assess the change in muscle thickness and echogenicity as markers of muscle quality, evaluated through ultrasonography in the tibialis anterior muscles of the lower limbs of participants undergoing 8 weeks of resistance training

Secondary objectives include:

* Characterize muscle architecture through ultrasonographic evaluation (fascicle length, pennation angle, and muscle thickness).
* Assessing changes in body composition.
* Evaluating muscle regeneration biomarkers.
* Determining the impact on respiratory muscle strength and aerobic capacity
* Evaluate maximal handgrip strength
* Assess overall lower-limb strength
* Assess overall upper-limb strength
* Measure maximal voluntary isometric strength
* Evaluate functional ankle muscle strength
* Determine maximal lower-limb muscle strength
* Assess balance and gait performance
* Evaluate health-related quality of life (HRQoL)
* Analyze body composition
* Investigate muscle regeneration
* Monitor physical activity levels

Materials and Methods: This clinical trial will recruit 22 participants (n=11 with HSPN, n=11 without HSPN), aged 15-29 years. Participants will be assigned to an 8-week supervised lower-limb RET program, performed 3 times per week, with progressive loads from 60% to 80% of one-repetition maximum (1RM). Exercises will target the major lower limb muscle groups and include leg press, knee extension, knee flexion, and ankle dorsiflexion.

Assessments will be conducted pre- and post-intervention, including:

* Muscle architecture and composition via ultrasound (tibialis anterior thickness, fascicle length, pennation angle, echogenicity).
* Muscle strength tests (isometric voluntary contraction, 1RM, grip strength).
* Functional capacity tests (6-minute walk test, balance assessment).
* Body composition (bioimpedance, anthropometry).
* Health-related quality of life (SF-36 questionnaire).
* Blood markers for muscle regeneration (creatine kinase). All participants will maintain habitual diet and physical activity levels during the intervention.

Expected Results: It is hypothesized that 8 weeks of progressive RET will result in greater improvements in muscle quality, functional capacity, and quality of life compared to baseline in both groups, with greater relative improvements expected in participants with HSPN due to lower baseline values. Increases in tibialis anterior thickness and reductions in echogenicity are expected, along with improvements in muscle strength, aerobic capacity, and balance. No serious adverse events are anticipated.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between 15 and 29 years of age with a diagnosis of hereditary sensorimotor polyneuropathy (HSPN) in any of its subtypes, living in the community (for experimental group).
* Healthy men or women between 15 and 29 years of age living in the community (for control group).
* Having active ankle movement within a range from plantarflexion to at least 0° of ankle dorsiflexion, allowing for strength training.

Exclusion Criteria:

* Osteoarticular or mobility impairments that prevent safe performance of resistance exercise training (e.g., ankle arthrodesis).
* Use of nutritional supplements that may affect skeletal muscle regulation (leucine, glutamine, casein, whey protein, fatty acids, creatine, among others).
* Untreated and/or uncontrolled chronic diseases or intellectual disability.
* History of surgery
* Participation in a resistance exercise training program within the past 6 months.

Ages: 15 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2026-07-20 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Changes in muscle echogenicity as marker of muscle quality | The evaluation will be conducted twice, before and after the 8-week intervention: the first, 2 days after signing the informed consent, and the second, 2 days after completing the treatment.
  .Echogenicity of the tibialis anterior muscle in both lower limbs will be assessed using ultrasonography (GE Logiq e BT11, 10-MHz linear transducer) by an experienced examiner. Participants will be seated with knees flexed and feet supported; the head of the fibula and lateral malleolus will serve as reference points. Echointensity will be analyzed in ImageJ from transverse images, excluding bone and fascia, and expressed as 0-255 A.U.
Changes in muscle thickness as marker of muscle quality | The evaluation will be conducted twice, before and after the 8-week intervention: the first, 2 days after signing the informed consent, and the second, 2 days after completing the treatment.
  Muscle thickness of the tibialis anterior muscle in both lower limbs will be assessed using ultrasonography (GE Logiq e BT11, 10-MHz linear transducer). Participants will be seated with knees flexed and feet supported; the head of the fibula and the lateral malleolus will serve as anatomical reference points.
  Muscle thickness will be defined as the orthogonal distance between the superficial and deep aponeuroses, measured at the midpoint of the transverse ultrasonographic image expressed in millimeters (mm).

SECONDARY OUTCOMES:
Changes in muscle architecture through ultrasonographic evaluation (fascicle length and pennation angle) | The evaluation will be conducted twice, before and after the 8-week intervention: the first, 2 days after signing the informed consent, and the second, 2 days after completing the treatment.
  Measurements will be performed on the tibialis anterior muscle of both lower limbs using ultrasonography (GE Logiq e BT11, General Electric, Boston, MA, USA) with a 10-MHz linear transducer by an evaluator experienced in muscle ultrasound analysis. For the assessment, participants will be positioned in a seated posture with knees flexed in neutral position and feet supported without footwear. The head of the fibula and the center of the lateral malleolus will be used as anatomical landmarks, where the total length will be measured and divided into three portions. Measurements will be obtained with the transducer placed transversely on the muscle belly located in the upper third of the distance measured between the two aforementioned bony landmarks. The analysis of muscle architecture will be performed using the public-domain software NIH ImageJ. This quantification will also be carried out by a blinded evaluator.
Serum creatine kinase concentration as a biomarker of muscle quality. | The evaluation will be conducted twice, before and after the 8-week intervention: the first, 2 days after signing the informed consent, and the second, 2 days after completing the treatment.
  Blood samples will be collected in the morning after a 12-hour fasting period from a superficial vein in the cubital fossa. Samples will be obtained on the first evaluation day (1 week before starting training) and 48 hours after the final training session. They will be drawn into serum-separator tubes without anticoagulant, centrifuged at 2500 rpm for 15 minutes, and the resulting serum will be aliquoted into microtubes and stored at -80 °C for subsequent analysis of Creatine Kinase levels.
Changes in total body mass | The evaluation will be conducted twice, before and after the 8-week intervention: the first, 4 days after signing the informed consent, and the second, 4 days after completing the treatment.
  Total and regional lean body mass will be assessed by bioelectrical impedance analysis (HBF-514C, Omron©, Japan) after overnight fasting, with participants standing. Lean body mass will be expressed in kilograms (kg) and as a percentage of total body mass (%).
Variation in anthropometric measurements | The evaluation will be conducted twice, before and after the 8-week intervention: the first, 4 days after signing the informed consent, and the second, 4 days after completing the treatment.
  anthropometric measurements will include body weight measured in kilograms (Kg), height, waist to hip, chest, thigh, and calf circumferences, as well as knee height and leg length mesuared in milimiters (mm). Weight and height will be obtained with a SECA® platform scale and stadiometer (Madison, WI, USA), while circumferences will be measured with a retractable SECA® measuring tape at standardized anatomical landmarks. Weight and height will be combined to report BMI in kg/m^2
Changes in aerobic capacity | The evaluation will be conducted twice, before and after the 8-week intervention: the first, 4 days after signing the informed consent, and the second, 4days after completing the treatment.
  Oxygen consumption (VO₂) will be measured during the 6-Minute Walk Test (6MWT) using a portable metabolic analyzer (PNOE, ENDO Medical, Palo Alto, CA). Breath-by-breath respiratory gas exchange kinetics will be recorded, while heart rate will be continuously monitored with an ECG-activated POLAR® chest strap (Finland). VO₂, VCO₂ and tidal volume, be assessed via a face mask equipped with a flow sensor and gas analyzer with minimal dead space (<70 ml). Data will be transmitted in real time to a laptop through a harness-secured system, enabling continuous monitoring throughout the tests.
Changes in respiratory muscle strength | The evaluation will be conducted twice, before and after the 8-week intervention: the first, 4 days after signing the informed consent, and the second, 4 days after completing the treatment.
  Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) will be assessed using a portable handheld spirometer (MicroRPM, Micro Medical/CareFusion, Kent, UK). Measured in centimeters of water (cmH₂O)
Changes in maximal handgrip strength | The evaluation will be conducted twice, before and after the 8-week intervention: the first, 2 days after signing the informed consent, and the second, 2 days after completing the treatment.
  Handgrip strength will be measured using a JAMAR dynamometer (model BK-7498, Fred Sammons, Inc., Burr Ridge, IL) for both upper limbs. Each hand will be tested three times with a 30-second rest between trials, and the highest value from the six attempts will be recorded
Changes in overall lower-limb strength | The evaluation will be conducted twice, before and after the 8-week intervention: the first, 2 days after signing the informed consent, and the second, 2 days after completing the treatment.
  This will be assessed using the Sit-to-Stand Test (STST). The participant will sit on a chair with arms crossed over the chest and, upon the command 'ready, go,' will stand up and sit down as many times as possible within 1 minute. The total number of repetitions will be recorded.
Changes in overall upper-limb strength | The evaluation will be conducted twice, before and after the 8-week intervention: the first, 2 days after signing the informed consent, and the second, 2 days after completing the treatment.
  Upper-limb strength will be assessed with the 30-s Arm Curl Test using a dumbbell (2.5 kg for women, 3.5 kg for men), recording the number of full elbow flexion-extension repetitions completed in 30 seconds
Changes in maximal voluntary isometric strength | The evaluation will be conducted twice, before and after the 8-week intervention: the first, 2 days after signing the informed consent, and the second, 2 days after completing the treatment.
  Maximal voluntary isometric strength of the ankle dorsiflexors will be assessed bilaterally using a force transducer (Load Cell -500 lb, Sensortronics, USA). After a 5-minute ankle mobility warm-up, participants will be seated with the trunk supported, hip at 90°, knee extended, and foot perpendicular to the transducer. The best of three maximal dorsiflexion trials, performed at high speed with verbal encouragement, will be recorded.
Changes in functional ankle muscle strength | The evaluation will be conducted twice, before and after the 8-week intervention: the first, 2 days after signing the informed consent, and the second, 2 days after completing the treatment.
  This will be assessed using the Heel Raise Test. The participant will stand facing a platform or step, keeping the body upright and feet parallel with the forefoot placed on the platform edge, while supporting themselves on the wall with both hands. They will be instructed to rise onto the toes as many times as possible within 30 seconds, and the total number of repetitions will be recorded.
Changes maximal lower-limb muscle strength | The evaluation will be conducted twice, before and after the 8-week intervention: the first, 2 days after signing the informed consent, and the second, 2 days after completing the treatment.
  Maximal strength will be determined through a one-repetition maximum (1RM) test for the lower limbs using leg press and knee extension machines (TuffStuff Fitness International), as well as free weights for ankle dorsiflexion and plantarflexion exercises
Changes in balance and gait performance | The evaluation will be conducted twice, before and after the 8-week intervention: the first, 4 days after signing the informed consent, and the second, 4 days after completing the treatment.
  Blance and Gait will be assessed with the Tinetti Performance-Oriented Mobility Assessment (POMA), which includes 22 items divided into gait (12 points) and balance (16 points), for a total of 28 points. Scores of 19-24 indicate minimal fall risk, while scores <19 indicate high fall risk.
Changes in health-related quality of life (HRQoL) | The evaluation will be conducted twice, before and after the 8-week intervention: the first, 4 days after signing the informed consent, and the second, 4 days after completing the treatment.
  Health-related quality of life will be assessed with the SF-36, a validated 36-item questionnaire covering 8 domains and 2 summary components (Physical Component Summary and Mental Component Summary). Scores range from 0 to 100%, with higher scores indicating better quality of life.
Changes physical activity levels | The evaluation will be conducted twice, before and after the 8-week intervention: the first, 4 days after signing the informed consent, and the second, 4 days after completing the treatment.
  The International Physical Activity Questionnaire (IPAQ) assesses physical activity levels across four domains: work, domestic, transport, and leisure time. Physical activity is expressed both continuously, in metabolic equivalent (MET)-minutes/week, and categorically, classifying activity level as low, moderate, or high. METs provide a way to estimate energy expenditure as multiples of basal metabolic rate, and the unit used, MET-minutes, is calculated by multiplying the MET value of an activity by the minutes performed per day or per week. In this study, results will be expressed in MET-minutes/week.

CONTACTS AND LOCATIONS:
Locations (2):
- Chile (2):
  - Temuco, Chile, Temuco, La Araucanía
  - Universidad de La Frontera, Temuco, La Araucanía

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be shared due to ethical restrictions and the risk of participant re-identification, as the informed consent did not include provisions for public data sharing.

REFERENCES:
- See also: The American College of Sports Medicine (ACSM) is a leading global organization dedicated to advancing and integrating scientific research, education, and practical applications in sports medicine, exercise science, and physical activity. — https://acsm.org/